CLINICAL TRIAL: NCT00343785
Title: Cyclophosphamide and Antithymocyte Globulin Conditioning Regimen for Marrow Transplantation From HLA-Matched Family Members for Severe Aplastic Anemia: Effect of Marrow Cell Dose on Chronic Graft-vs.-Host Disease: A Multi-Center Trial
Brief Title: Cyclophosphamide and Anti-thymocyte Globulin Followed By Methotrexate and Cyclosporine in Preventing Chronic Graft-Versus-Host Disease in Patients With Severe Aplastic Anemia Undergoing Donor Bone Marrow Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Rainer Storb, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2054.00; NCI-2010-01781 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P01HL036444 (NIH)
Record Dates: First submitted 2006-06-22; First posted 2006-06-23 (Estimated); Results first posted 2017-03-16 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-03

CONDITIONS: Aplastic Anemia
MeSH Terms: conditions — Anemia, Aplastic | interventions — Cyclophosphamide; Antilymphocyte Serum; thymoglobulin; Cyclosporine; Transplantation; Methotrexate; merphos; Flow Cytometry; Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (conditioning regimen, transplant, GVHD prophylaxis) (Experimental): Patients receive a conditioning regimen comprising cyclophosphamide IV on days -5 to -2 and anti-thymocyte globulin IV over 4-10 hours on days -4 to -2. Patients undergo allogeneic bone marrow transplantation on day 0. Patients then receive GVHD prophylaxis comprising methotrexate IV on days 1, 3, 6, and 11 and cyclosporine IV over 1 hour or PO twice daily on days -1 to 50, followed by a taper until 6 months after grafting.
  Interventions: Drug: cyclophosphamide; Biological: anti-thymocyte globulin; Drug: cyclosporine; Procedure: allogeneic bone marrow transplantation; Drug: methotrexate; Genetic: DNA analysis; Other: flow cytometry; Genetic: polymorphism analysis; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Biological: anti-thymocyte globulin — Given IV
  Other Names: ATG; ATGAM; lymphocyte immune globulin; Thymoglobulin
Drug: cyclosporine — Given IV or PO
  Other Names: ciclosporin; cyclosporin; cyclosporin A; CYSP; Sandimmune
Procedure: allogeneic bone marrow transplantation — Undergo allogeneic bone marrow transplantation
  Other Names: bone marrow therapy, allogeneic; bone marrow therapy, allogenic; transplantation, allogeneic bone marrow; transplantation, allogenic bone marrow
Drug: methotrexate — Given IV
  Other Names: amethopterin; Folex; methylaminopterin; Mexate; MTX
Genetic: DNA analysis — Correlative studies
Other: flow cytometry — Correlative studies
Genetic: polymorphism analysis — Correlative studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This clinical trial is studying how well giving cyclophosphamide together with anti-thymocyte globulin followed by methotrexate and cyclosporine works in preventing chronic graft-vs-host disease (GVHD) in patients with severe aplastic anemia undergoing donor bone marrow transplant. Giving low doses of chemotherapy, such as cyclophosphamide, before a donor bone marrow transplant helps stop the growth of abnormal cells. It also stops the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune system and help destroy any remaining abnormal cells. Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving anti-thymocyte globulin before and methotrexate and cyclosporine after transplant may stop this from happening

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Minimize the incidence of chronic GVHD by restricting the transplanted marrow dose to 2.0-2.5 x 10^8 nucleated cells/kg.

SECONDARY OBJECTIVES:

I. Engraftment and overall survival.

OUTLINE:

CONDITIONING REGIMEN: Patients receive cyclophosphamide intravenously (IV) on days -5 to -2 and anti-thymocyte globulin IV over 4-10 hours on days -4 to -2.

TRANSPLANTATION: Patients undergo allogeneic bone marrow transplantation on day 0.

GVHD PROPHYLAXIS: Patients receive methotrexate IV on days 1, 3, 6, and 11 and cyclosporine IV over 1 hour or orally (PO) twice daily on days -1 to 50, followed by a taper until 6 months after grafting.

After completion of study treatment, patients are followed up at on day 180, 1 year, 1.5 years, 2 years, 3 years, and yearly thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who has aplastic anemia with marrow failure involving 2 of the three following criteria: granulocytes < 500/uL; a corrected reticulocyte count of < 1%; platelet count of < 20,000/uL
* Availability of an human leukocyte antigen (HLA)-matched family member
* DONOR: Family member who is HLA-matched
* DONOR: If more than one HLA-matched family member is available, priority will be given to a donor who is genotypically HLA-identical, of appropriate cytomegalovirus (CMV) serology, ABO compatible, and, in case of a female donor, non-parous

Exclusion Criteria:

* Severe disease other than aplastic anemia that would severely limit the probability of survival during the graft procedure:

  * Patients who have developed clonal cytogenetic abnormalities or myelodysplastic syndrome (preleukemia)
  * Patients with Fanconi's anemia
  * Aplasia secondary to radiation or cytotoxic chemotherapy
  * Patients with paroxysmal nocturnal hemoglobinuria who have not developed aplastic anemia
* Severe organ toxicities:

  * Cardiac insufficiency requiring treatment or symptomatic coronary artery disease;
  * Severe hypoxemia , partial pressure of oxygen (pO2) < 70 mm Hg, with decreased diffusion capacity of carbon monoxide (DLCO) < 70% of predicted; or mild hypoxemia, pO2 < 80 mm Hg with severely decreased DLCO < 60% of predicted;
  * Impaired renal function (creatinine > 2 times upper limit of normal or estimated creatinine clearance < 60 ml/min)
* Fungal infections with radiological progression after receipt of amphotericin B or active triazole for greater than 1 month
* Human immunodeficiency virus (HIV)-positive patients
* Females who are pregnant or breast-feeding
* DONOR: Donors who have increase anesthetic risk and are not able psychologically and medically to tolerate the procedure
* DONOR: HIV-positive donors

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2006-02; Primary Completion 2012-05 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Storb, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (3):
- United States (3):
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Conditioning Regimen, Transplant, GVHD Prophylaxis)
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Conditioning Regimen, Transplant, GVHD Prophylaxis)
Number analyzed (Participants) | 21
Age, Continuous [Median (Full Range); unit: years] | 15 [3 to 52]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 3
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Chronic GVHD
Description: Analyzed using cumulative incidence estimates, treating death or rejection as competing risk events.
Time Frame: 2 years
Population: All Patients
Measure: Number; unit: number participants with chronic GVHD
Groups:
- Patients Receive a Conditioning Regimen Comprising Cyclophosph: Patients receive a conditioning regimen comprising cyclophosphamide IV on days -5 to -2 and anti-thymocyte globulin IV over 4-10 hours on days -4 to -2. Patients undergo allogeneic bone marrow transplantation on day 0. Patients then receive GVHD prophylaxis comprising methotrexate IV on days 1, 3, 6, and 11 and cyclosporine IV over 1 hour or PO twice daily on days -1 to 50, followed by a taper until 6 months after grafting.
Arm/Group | Patients Receive a Conditioning Regimen Comprising Cyclophosph
Number analyzed (Participants) | 21
number participants with chronic GVHD | 5

2. Secondary Outcome: Number of Days to Neutrophil Recovery to >500/uL
Description: First of 3 consecutive days of neutrophils >500/uL
Time Frame: 100 days post-transplant
Population: All patients
Measure: Median (Full Range); unit: days
Arm/Group | Treatment (Conditioning Regimen, Transplant, GVHD Prophylaxis)
Number analyzed (Participants) | 21
days | 26 [21 to 36]

3. Secondary Outcome: Overall Survival
Description: Number of patients alive at one year
Time Frame: From the time of enrollment until death from any cause up to one year
Population: All Patients
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Conditioning Regimen, Transplant, GVHD Prophylaxis)
Number analyzed (Participants) | 21
Participants | 21

ADVERSE EVENTS:
Arm/Group | Treatment (Conditioning Regimen, Transplant, GVHD Prophylaxis)
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 5/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Conditioning Regimen, Transplant, GVHD Prophylaxis) (N=21)
parental nutrition (Gastrointestinal disorders) | 3 (3) — mucositis requiring parental nutrition
hypertension (Cardiac disorders) | 2 (2)
hyperbilirubinemia (Hepatobiliary disorders) | 1 (1) — bilirubin > 3x ULN, cholangitis lenta
Tinnitus (Ear and labyrinth disorders) | 1 (1) — significant tinnitus in both ears with hearing loss, correctable with hearing aids
hypoxia (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Conditioning Regimen, Transplant, GVHD Prophylaxis) (N=21)
nausea (Gastrointestinal disorders) | 21 (21)
vomiting (Gastrointestinal disorders) | 21 (21)
mucositits (Gastrointestinal disorders) | 21 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes